CLINICAL TRIAL: NCT00478491
Title: fMRI of Vulnerable Brain Regions in Persons at Risk for Alzheimer's Disease
Acronym: ALZ
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2002-515; NIH RO1 AG021155A
Record Dates: First submitted 2007-05-22; First posted 2007-05-24 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Magnetic Resonance Imaging; Alzheimer's Disease; Dementia; Adult Children; Risk
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma and serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- 1: Persons with a parent with Alzheimer's disease
- 2: Persons whose parents survived to old age without memory problems
- 3: Persons with diagnosed mild cognitive impairment
- 4: Persons without memory problems

SUMMARY:
The purpose of this study is to investigate the organization of memory and develop future methods for early detection of AD. Using functional magnetic resonance imaging (fMRI), we examine the responsiveness of the brain to memory tasks, specifically focusing on regions of the brain (the mesial temporal lobe and posterior cingulate) that are known to be involved in early stages of Alzheimer's disease (AD). Of interest are differences in brain activation between people with and without a family history of AD and other risk factors.

ELIGIBILITY:
Inclusion Criteria:

* MCI Group: Diagnosis of mild cognitive impairment
* AD Family History Group: Confirmed family history of Alzheimer's and concurrent enrollment in the Wisconsin Registry for Alzheimer's Prevention (WRAP)
* Control Groups: Cognitively healthy and both parents survived past age 70 with no memory problems

Exclusion Criteria:

* Claustrophobia
* Metallic or electronic implants or devices that are not MRI-safe

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Persons with a parent with Alzheimer's disease will be recruited from the Wisconsin Registry for Alzheimer's Prevention (WRAP). Persons with MCI will be recruited from the UW clinics and satellite clinics. Controls for the above study groups will be recruited from the WRAP and the local community.
Sampling Method: Non-Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2003-01; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sterling C Johnson, PhD, Principal Investigator — University of Wisconsin/VA GRECC
Locations (1):
- University of Wisconsin - Wisconsin Comprehensive Memory Program, Madison, Wisconsin, United States

REFERENCES:
- [Result] Ries ML, Jabbar BM, Schmitz TW, Trivedi MA, Gleason CE, Carlsson CM, Rowley HA, Asthana S, Johnson SC. Anosognosia in mild cognitive impairment: Relationship to activation of cortical midline structures involved in self-appraisal. J Int Neuropsychol Soc. 2007 May;13(3):450-61. doi: 10.1017/S1355617707070488. PMID 17445294
- [Result] Johnson SC, Schmitz TW, Trivedi MA, Ries ML, Torgerson BM, Carlsson CM, Asthana S, Hermann BP, Sager MA. The influence of Alzheimer disease family history and apolipoprotein E epsilon4 on mesial temporal lobe activation. J Neurosci. 2006 May 31;26(22):6069-76. doi: 10.1523/JNEUROSCI.0959-06.2006. PMID 16738250
- [Result] Trivedi MA, Schmitz TW, Ries ML, Torgerson BM, Sager MA, Hermann BP, Asthana S, Johnson SC. Reduced hippocampal activation during episodic encoding in middle-aged individuals at genetic risk of Alzheimer's disease: a cross-sectional study. BMC Med. 2006 Jan 13;4:1. doi: 10.1186/1741-7015-4-1. PMID 16412236
- [Result] Ward MA, Carlsson CM, Trivedi MA, Sager MA, Johnson SC. The effect of body mass index on global brain volume in middle-aged adults: a cross sectional study. BMC Neurol. 2005 Dec 2;5:23. doi: 10.1186/1471-2377-5-23. PMID 16321166
- [Result] Ries ML, Schmitz TW, Kawahara TN, Torgerson BM, Trivedi MA, Johnson SC. Task-dependent posterior cingulate activation in mild cognitive impairment. Neuroimage. 2006 Jan 15;29(2):485-92. doi: 10.1016/j.neuroimage.2005.07.030. Epub 2005 Aug 15. PMID 16102979
- See also: Website for the Sterling Johnson Imaging Lab — http://www.brainmap.wisc.edu